CLINICAL TRIAL: NCT04963608
Title: Real World Study of Inetetamab HER2 Positive Advanced Breast Cancer
Brief Title: RWS of Inetetamab HER2 Positive Advanced Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhiyong Yu (Other)
Responsible Party: Sponsor-Investigator, Zhiyong Yu, Chief of breast department, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Other Study IDs: RSINETE
Record Dates: First submitted 2021-07-11; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: HER2-positive Advanced Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- non-interventional study: Her2 positive ABC patients who have received Inetetamab in the metastatic setting.
  Interventions: Drug: Inetetamab

INTERVENTIONS:
Drug: Inetetamab — 8mg/kg iv day 1 followed by 6mg/kg iv day 1, cycled every 21 days

SUMMARY:
This non-Interventional study will describe and analyze the clinical use of Inetetamab in clinical practice in the treatment of HER2 positive advanced breast cancer in the real world.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stage IV breast cancer
2. Patients with HER2 positive status
3. Patients that received Inetetamab
4. Patients that began Inetetamab therapy prior to June 30, 2021.

Exclusion Criteria:

Patients treated with an investigational anticancer agent Inetetamab

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER2+ advanced breast cancer patients whose treatment decision with Inetetamab has been made by their physician and who meet the eligibility criteria will be invited to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival(PFS) | 12 months
Incidences of adverse events and toxicities | 12 months

IPD SHARING:
Plan to Share IPD: Undecided
The results of this retrospective observational study will not be formally documented in a Clinical Study Report. Coded patient-level data will be shared with the sponsor.